CLINICAL TRIAL: NCT06823206
Title: Effects of Movement Representation Techniques with Sensorimotor Training for Rotator Cuff Related Shoulder Pain: a Randomised Controlled Trial
Brief Title: Effects of Movement Representation Techniques with Sensorimotor Training for Rotator Cuff Related Shoulder Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, LEONG Hio Teng Annie, Principal Investigator, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20231205001
Record Dates: First submitted 2025-01-09; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Rotator Cuff Related Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Wait-list control
- Intervention (Experimental)
  Interventions: Other: Sensorimotor training with movement representation techniques

INTERVENTIONS:
Other: Sensorimotor training with movement representation techniques — Sensorimotor training will be implemented with movement representation techniques using a standardized retraining sequence of a shoulder control exercise during arm elevation with 3 phases: Phase 1: Action Observation Training; Phase 2: Mirror therapy; and Phase 3: Sensorimotor training of the involved arm. Each session will last 60 minutes, with one supervised intervention session over the 12 weeks.
  Arms: Intervention

SUMMARY:
The aim of this study is to evaluate the efficacy of 12 weeks of sensorimotor training with movement representation techniques for reducing pain intensity in people with rotator cuff related shoulder pain, relative to standard care. Besides, the secondary aim of this study is to explore the mechanisms underlying the effects of central mechanism treatment in people with rotator cuff related shoulder pain. A total of 122 older adults aged 50 or above with the presence of shoulder pain for more than three months will be recruited and randomized into 12-weeks of movement representation techniques with sensorimotor training vs. standard care. Shoulder pain and disability Index (SPADI), changes in primary motor cortex (M1) using brain MRI, changes in subacromial space using ultrasound imaging, Widespread Pain Index (WPI), Pain Catastrophising Scale (PCS), and Fear-avoidance Beliefs questionnaires (FABQ) will be assessed at baseline and 12-week post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 or above
* Presence of shoulder pain for more than three months
* Clinical test showed 3/5 positive tests (painful arc, resisted external rotation, Neer test, Kennedy-Hawkins test, and Jobe test), and the intensity of pain being provoked should be ≥ 3/10 on an 11-point numeric pain rating scale (NPRS)
* Structural changes of rotator cuff tendons using MRI or ultrasound imaging

Exclusion Criteria:

* History of trauma
* Shoulder fracture, glenohumeral osteoarthritis, or arthritis in the acromioclavicular joint
* Clinically suspected labrum lesion
* Previous shoulder surgery or dislocation
* Clinical signs of anterior shoulder instability
* Clinical signs of frozen shoulders
* Previous clinical treatment or corticosteroid injection for a shoulder injury within the last 12 months
* Symptoms referred from or related to the spine; and (9) other competing diagnoses (i.e., rheumatoid arthritis, cancer, neurological disorders, fibromyalgia, or psychiatric illness).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline and 12-weeks post-intervention
  Pain will be assessed using the pain sub-score of the Chinese Version of the Shoulder Pain and Disability Index. It is a validated self-administered questionnaire used to evaluate upper limb symptoms and functional limitations during daily activities. The questionnaire consists of 13 items with two subscales, i.e., pain intensity (five items) and disability (eight items), and each subscale-item will be summed to obtain a pain-score and a disability-score. The total of all items will be summed to obtain the final scores for each domain ranging from 0 to 100, with higher scores indicating more pain and disability. In the present study, the pain sub-score will be used as the measure of average pain intensity.

SECONDARY OUTCOMES:
Cortical thickness in the primary motor cortex (M1) using brain MRI | Baseline and 12 weeks post-intervention
  The brain structure will be measured using structural and resting-state functional magnetic resonance imaging (fMRI) on a 3.0 T Siemens Prisma scanner. During the resting-state scan, the participants will be instructed to rest with their eyes closed while remaining stationary for 30 minutes. The regional cortical thickness of the brain region, the primary motor cortex (M1), will be extracted from T1-weighted MRI images.

OTHER OUTCOMES:
Shoulder strength | Baseline and 12-weeks post-intervention
  The isokinetic testing of shoulder rotational strength will be measured using a Cybex Norm isokinetic dynamometer
Subacromial space | Baseline and 12-weeks post-intervention
  The subacromial space will be scanned using an ultrasound scanning system during arm resting at 0° and static arm holding at 60° of shoulder abduction. The subacromial space will be measured from the tangential distance between the humeral head and the infero-lateral edge of the acromion. Three measurements will be recorded and the averaged value will be calculated.
Central pain processing | Baseline and 12-weeks post-intervention
  The Widespread Pain Index will be adopted to capture features of central sensitisation. It quantifies the extent of bodily pain on a 0-19 scale, assessing whether patients have pain in 19 different body regions, each point scores 1. All items will be summed to obtain a final score ranging from 0 to 100, with higher scores indicating more widespread pain.
Pain Catastrophising | Baseline and 12-weeks post-intervention
  The Chinese version of the Pain Catastrophising Scale will be used to assess pain catastrophising. This is a validated self-administered questionnaire consisting of 13-items examining pain-related behaviours and cognition. Scores range from 0 to 52, with higher scores indicating a higher level of catastrophising.
Fear-avoidance Beliefs questionnaires | Baseline and 12-weeks post-intervention
  The Chinese version of the Fear-avoidance Beliefs questionnaires is a self-administered questionnaire consisting of 16 items with 2 subscales that evaluate fear avoidance beliefs about physical activity and work. Each item is scored from 0 to 6, representing completely disagree to completely agree. The total score is calculated by the summation of the individual scores of each item, from 0 to 96, with higher scores indicating a higher degree of fear avoidance belief.

IPD SHARING:
Plan to Share IPD: Undecided